CLINICAL TRIAL: NCT04061239
Title: Primary Comparison of Liposomal Anthracycline Based Treatment Versus Conventional Care Strategies Before Allogeneic Stem Cell Transplantation in Patients With Higher Risk MDS and Oligoblastic AML
Brief Title: Comparison of Therapies Before Stem Cell Transplantation in Patients With Higher Risk MDS and Oligoblastic AML
Acronym: PALOMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALOMA
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: MDS; AML
MeSH Terms: interventions — CPX-351; Daunorubicin; Cytarabine; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPX-351 Arm (Experimental): CPX-351 is a liposomal formulation with a fixed 5:1 molar ratio of cytarabine and daunorubicin. It will be administered as a 90-minute intravenous infusion.
  The treatment includes up to 2 cycles of induction as follows:
  * 1 x CPX-351 1st induction: daunorubicin 44 mg/m² and cytarabine 100 mg/m² in liposomes on days 1, 3, and 5
  * 1 x CPX-351 2nd induction: daunorubicin 44 mg/m² and cytarabine 100 mg/m² in liposomes on days 1 and 3
  Each induction cycle will last 28 days. Depending on the type and extent of response as well as toxicity, the patient may continue on to consolidation therapy after induction or be discontinued from the treatment phase and transferred directly to alloHCT, if applicable. CPX-351 consolidation is with daunorubicin 29 mg/m² and cytarabine 65 mg/m² in liposomes on days 1 and 3. For patients < 60 years up to 3 consolidation cycles and for patients ≥ 60 years up to 2 consolidation cycles are allowed.
  Interventions: Drug: CPX-351
- CCR Arm (Other): The conventional care regimens (CCR) arm has 2 options according to the discretion of the investigator:
  1. conventional "7+3" cytarabine/daunorubicin chemotherapy regimen
  2. treatment with s.c. Azacitidine
  Interventions: Drug: Daunorubicin; Drug: Cytarabine; Drug: Azacitidine

INTERVENTIONS:
Drug: CPX-351 — CPX-351 is a liposomal formulation with a fixed 5:1 molar ratio of cytarabine and daunorubicin. It will be administered as a 90-minute intravenous infusion.
  Other Names: Vyxeos
  Arms: CPX-351 Arm
Drug: Daunorubicin — Daunorubicin is commercially available as a powder for reconstitution in 20 mg vials. In this trial, daunorubicin should be administered as an IV infusion over 60 min.
  Arms: CCR Arm
Drug: Cytarabine — Cytarabine is commercially available as vials/bottles for preparation of diluted infusion solution. Cytarabine will be administrated intravenously. In this trial, cytarabine is administered as a continuous infusion.
  Arms: CCR Arm
Drug: Azacitidine — Azacitidine at 75mg/m² for 7 days. Patients should receive a minimum of 2 and up to 6 cycles.
  Other Names: Vidaza
  Arms: CCR Arm

SUMMARY:
To compare the event-free survival at 2 years of CPX-351 vs. conventional care regimens before allogeneic blood cell transplantation as first line treatment in patients with higher risk MDS and oligoblastic AML.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (alloHCT) is considered the only potentially curative treatment option for MDS patients and is therefore often considered the standard treatment for mainly higher-risk MDS patients up to the age of 75 years. One common approach to "bridge" higher-risk MDS from the time of diagnosis to transplantation is a treatment with hypomethylating agents such as azacitidine due to its anticipated low toxicity profile. Alternative strategies are intensive 7+3 chemotherapy with anthracycline and cytarabine or direct and immediate transplantation. By this strategy the time interval for donor search can be significantly prolonged leading to a higher proportion of success.Nevertheless, not every patient initially eligible for transplantation undergoes this procedure subsequently. A direct prospective comparison of different therapeutic approaches as outlined above versus CPX-351 prior to alloHCT has not been performed so far and is subject of the PALOMA trial. We hypothesize that CPX-351 will lead to higher and more durable response rates including a more favourable safety profile and long-term outcome compared to currently used conventional care regimens approaches prior to alloHCT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients, 18-75 years of age
* Diagnosis of high risk MDS including oligoblastic non-proliferative (WBC <13 Gpt/l) AML up to 29% of bone marrow blasts
* Availability of BM blast count from central morphology
* Bone marrow blasts ≥ 5%
* IPSS score intermediate or high
* alloHCT intended within the next 6 months
* ECOG performance status of 0 or 1
* Signed informed consent
* Laboratory values fulfilling the following:
* Serum creatinine < 2.0 mg/dL
* Serum total bilirubin < 2.0 mg/dL
* Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN
* Cardiac ejection fraction (LVEF) ≥ 50% by echocardiography
* Contraception:
* Female subjects of childbearing potential† must agree to use a medically acceptable method of contraception for at least 2 months prior to the first dose of CPX-351 and consent of female patients to use a medically acceptable method of contraception throughout the entire study period and for 6 months following the last dose of CPX-351. Medically acceptable methods of contraception that may be used by the patient include abstinence, diaphragm and spermicide, intrauterine device (IUD), condom and vaginal spermicide, hormonal contraceptives (patients must be stable on hormonal contraceptives for at least the prior 3 months), surgical sterilization, or post-menopausal (≥2 years of amenorrhea). Medically acceptable methods of contraception that may be used by the male partner of a female patient are condom and spermicide or vasectomy (>6 months prior to Day-1) and are to be used throughout the entire study period and for 6 months following the last dose of CPX-351.
* Male patients must be willing to refrain from sperm donation for 6 months following the last dose of CPX-351 and must use adequate contraception throughout the entire study period and for 6 months following the last dose of CPX-351.
* Combined oral contraceptive pills are not recommended. It is recommended that during the study two medically accepted methods of contraception (e.g. as hormonal contraceptive methods along with a condom) apply.

Exclusion Criteria:

* Patients with history of myeloproliferative neoplasms (MPN) (defined as a history of essential thrombocytosis or
* polycythemia vera, or idiopathic myelofibrosis prior to the diagnosis of AML) or combined MDS/MPN are not eligible.
* WHO-2016 defined AML entities: AML with t(15;17), PML-RARA; AML with t(8;21), RUNX1-RUNX1T1, AML with inv(16)/t(16;16), CBFβ-MYH11; AML with biallelic CEBPA mutation; AML with mutated FLT3 or NPM1.
* Clinical evidence of active CNS leukemia.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
* Any major surgery or radiation therapy within four weeks prior screening.
* Patients with prior treatment of either CPX-351, hypomethylating agents, cytarabine or intensive chemotherapy for high-risk MDS or AML.
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent.
* Patients with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (NYHA Class III or IV staging).
* Active or uncontrolled infection. Patients with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs.
* Current evidence of invasive fungal infection (blood or tissue culture); patients with recent fungal infection must have a subsequent negative cultures to be eligible; known HIV (new testing not required) or evidence of active hepatitis B or C infection (with rising transaminase values).
* Hypersensitivity to cytarabine, daunorubicin or liposomal products.
* History of Wilson's disease or other copper-metabolism disorder.
* Female patients who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
2-year EFS in both arms | 2 years
  To compare the event-free survival (EFS) at 2 years of CPX-351 vs. CCR before allogeneic blood cell transplantation (alloHCT) as first line treatment in patients with higher risk MDS and oligoblastic AML.

SECONDARY OUTCOMES:
Response rate | 2 years
  To compare best and overall response rate of CPX-351 vs. CCR according to AML-ELN and MDS-IWG criteria
Toxicity Assessment | 2 years
  To compare the safety and tolerability of CPX-351 vs. CCR measured by NCI CTCAE v5.0
Proportion of patients proceeding to alloHCT | 2 years
  To compare the effects of CPX-351 vs. CCR on the proportion of patients proceeding to alloHCT
Minimal residual disease | 2 years
  To compare the effect of CPX-351 vs. CCR on minimal residual disease which will be assessed at all times of bone marrow puncture
Patient's quality of life | 2 years
  To compare the effect of CPX-351 vs. CCR on the quality of life. It will be measured using the EORTC-QLQ30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof., Principal Investigator — Universitätsklinikum Leipzig AöR
Locations (28):
- Austria (2):
  - Ordensklinikum Linz Elisabethinen GmbH, Linz
  - Uniklinikum Salzburg - Landeskrankenhaus, Salzburg
- Germany (26):
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Helios Klinikum Berlin-Buch GmbH, Berlin
  - Universitätsklinikum Bonn (UKB), Bonn
  - Klinikum Chemnitz-gGmbH, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Koblenz
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Universitätsmedizin Rostock, Rostock
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm